CLINICAL TRIAL: NCT04855539
Title: Coronavirus Infectious Disease 2019: Ventilator Outcomes Using Artificial Intelligence, Chest Radiographs and Other Evidence-based Co-variates (COVID VOICE)
Brief Title: Coronavirus: Ventilator Outcomes Using Artificial Intelligence Chest Radiographs & Other Evidence-based Co-variates
Acronym: COVID VOICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 232823
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- wave 1
- wave 2

SUMMARY:
We will determine ventilator outcomes to Coronavirus Infectious Disease 2019 (COVID-19) using artificial Intelligence with inputs of chest radiographs and other evidence-based co-variates.

DETAILED DESCRIPTION:
The chest radiograph (chest x-ray) has emerged as the United Kingdom's National Health Service (NHS) frontline diagnostic imaging test for COVID-19, in conjunction with clinical history and key blood markers: C-reactive protein (CRP) and lymphopenia. Typically, every suspected COVID-19 patient presenting to the emergency department is undergoing blood tests and a chest radiograph. Therefore, it has become critical for radiologists to review and "hot" report the chest x-ray urgently.

Primary Objective: Use chest radiographs and clinical data to determine whether patient can survive with a ventilator

ELIGIBILITY:
Inclusion Criteria:

Admitted to intensive care unit (ITU) or equivalent COVID-19 polymerase chain reaction (PCR) positive

Exclusion Criteria:

No imaging prior to ITU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults with COVID-19 at secondary and tertiary centres
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of a convolutional neural network to predict survival outcome | 1 month
  Defined by sensitivity, specificity, positive and negative predictive values

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Princess Royal University Hospital, Orpington, Kent
  - Guy's and St Thomas' Hospital, London
  - King's College Hospital, London